CLINICAL TRIAL: NCT00467688
Title: The Effect of Continuous Glucose Monitoring With and Without Real Time Access to Glucose Values and Glucose Alerts on Course of Glucose and Satisfaction With CGMS in Type 1 Diabetic Patients
Brief Title: Effect of Continuous Glucose Monitoring on Course of Glucose in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FIDAM 049-06; Nr.70-005928713-0
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: type 1 diabetes; glucose excursion; hypoglycemia awareness; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A,1 (No Intervention): Real time access to current measured glucose values; hyperglycemic or hypoglycemic alerts
  Interventions: Device: Real time access to current glucose values during CGMS
- A,2 (No Intervention): Retrospective analysis of glucose values
  Interventions: Device: Real time access to current glucose values during CGMS

INTERVENTIONS:
Device: Real time access to current glucose values during CGMS — One arm gets real time access to current measured glucose values and hypoglycemic or hyperglycemic alerts are elicited, The second arm get´s a retrospective analysis of glucose values

SUMMARY:
The objective of this cross over study is to access if continuous glucose monitoring (CGMS) with a real time feed back and hypoglycemic as well as hyperglycemic glucose alerts vs. only retrospective analysis of glucose values is able to improve course of glucose with special regard to time spent in hypoglycemic glucose ranges in type 1 diabetic patients with impaired hypoglycemia awareness or a history of severe hypoglycemia. The second objective is to access satisfaction with CGMS during both conditions

DETAILED DESCRIPTION:
The objective of this cross over study is to access if continuous glucose monitoring (CGMS) with a real time feed back and hypoglycemic as well as hyperglycemic glucose alerts vs. only retrospective analysis of glucose values is able to improve course of glucose with special regard to time spent in hypoglycemic glucose ranges. The second objective is to access satisfaction with CGMS during both conditions.

This study is conducted in an inpatient setting with type 1 diabetic patients. Partisans are asked to have twice a continuous glucose measurement with the GlucoDay System (Menarini Diagnostics). Each measurement period is limited to maximal 48 hours. In one condition the have real time access to current glucose values and alerts are given if glucose is dropping below 70 mg/dl or exceeding 180 mg/dl. During the other condition the participants are blind against their current glucose values and no alerts are given. Glucose course is retrospectively analyzed.

The order of these two conditions is randomized.

Expected outcome:

The primary outcome variable is the daily time spent in hypoglycemic range in type 1 diabetic patients with and without impaired hypoglycemia awareness or a history of severe hypoglycemia. Additionally the patients will also complete questionnaire about satisfaction with CGMS, diabetes related distress, treatment satisfaction, depressive and anxiety symptoms which belongs to the secondary variables.

Inclusion criteria:

* Type 1 diabetes
* Age > 18 years
* Informed consent

Exclusion criteria:

* Diagnosis and/or treatment of a current psychiatric disease
* Severe late complications

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Diagnosis and/or treatment of a current psychiatric disease
* Severe late complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Daily time spent in the hypoglycemic glucose range during continuous glucose measurement with and without real time access to glucose values and glucose alarms | during the 48 hours of using blind vs. unblind continuous glucose monitoring

SECONDARY OUTCOMES:
Time spent in euglycemic and hyperglycemic glucose range Satisfaction with CGMS Diabetes related distress Treatment satisfaction Anxiety and depressive symptoms | During and after the 48 hours measurement of CGMS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Haak, MD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim
Locations (2):
- Germany (2):
  - FIDAM, Bad Mergentheim
  - Research Institute of the Diabetes Academy Mergentheim, Bad Mergentheim

REFERENCES:
- [Derived] Hermanns N, Kulzer B, Gulde C, Eberle H, Pradler E, Patzelt-Bath A, Haak T. Short-term effects on patient satisfaction of continuous glucose monitoring with the GlucoDay with real-time and retrospective access to glucose values: a crossover study. Diabetes Technol Ther. 2009 May;11(5):275-81. doi: 10.1089/dia.2008.0078. PMID 19425875